CLINICAL TRIAL: NCT05359419
Title: Safety and Efficacy of Photodynamic Therapy With Aminolevulinic Acid 10% Topical Gel Activated by Red Light Versus Aminolevulinic Acid 20% Topical Solution Activated by Blue Light for the Treatment of Actinic Keratosis on the Upper Extremities: A Blinded Randomized Study
Brief Title: Comparison of Two Modes of Photodynamic Therapy for the Treatment of Actinic Keratosis on the Upper Extremities
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amezluz vs Levulan IIT 2022
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Ameluz (Experimental): AMELUZ® (aminolevulinic acid hydrochloride) gel, 10% with its approved light source (BF-RhodoLED® lamp, 635 nm ± 9 nm, Biofrontera, Inc., Wakefield, MA, US)
  Interventions: Combination Product: aminolevulinic acid hydrochloride gel, 10%
- Levulan (Active Comparator): LEVULAN® KERASTICK® (aminolevulinic acid HCl) topical solution, 20% with its approved light source (BLU-U® Blue light photodynamic Therapy Illuminator Model 4170, 417 nm ± 5 nm, DUSA Pharmaceuticals, Wilmington MA, US)
  Interventions: Combination Product: aminolevulinic acid HCl topical solution, 20%

INTERVENTIONS:
Combination Product: aminolevulinic acid hydrochloride gel, 10% — 10% ALA with Red Light
  Arms: Ameluz
Combination Product: aminolevulinic acid HCl topical solution, 20% — 20% ALA with Blue Light
  Arms: Levulan

SUMMARY:
This study will be a prospective clinical trial performed in a single center, with 20 adult subjects presenting 4-17 clinically confirmed, mild to moderate AKs according to Olsen grading on each of two comparable treatment fields on the hands and/or arms of the patients. Subjects will be randomize to receive treatment on one side with AMELUZ® (aminolevulinic acid hydrochloride) gel, 10% with its approved light source (BF-RhodoLED® lamp, 635 nm ± 9 nm, Biofrontera, Inc., Wakefield, MA, US) and the other side with LEVULAN® KERASTICK® (aminolevulinic acid HCl) topical solution, 20% with its approved light source (BLU-U® Blue light photodynamic Therapy Illuminator Model 4170, 417 nm ± 5 nm, DUSA Pharmaceuticals, Wilmington MA, US).

DETAILED DESCRIPTION:
This study will be a prospective clinical trial performed in a single center, with 20 adult subjects presenting 4-17 clinically confirmed, mild to moderate AKs according to Olsen grading on each of two comparable treatment fields on the hands and/or arms of the patients. The location and maximal size of the treatment fields should be such that PDT is possible with one illumination with BF-RhodoLED® and Blu-U® in parallel. The number of lesions on the two sides of a patient will not be allowed to differ by more than 50%.

Subjects will be treated on the AMELUZ® side according to the European SmPC with the exception that thea second PDT, if req uired, will be performed after two months (SmPC: three months), and on the LEVULAN® side according to the USPI. Subjects will be randomized as to which upper extremity (i.e. right vs. left) will receive AMELUZ® (aminolevulinic acid hydrochloride) gel, 10% with its approved light source (BF-RhodoLED® lamp, 635 nm ± 9 nm, Biofrontera, Inc., Wakefield, MA, US) or LEVULAN® KERASTICK® (aminolevulinic acid HCl) topical solution, 20% with its approved light source (BLU-U® Blue light photodynamic Therapy Illuminator Model 4170, 417 nm ± 5 nm, DUSA Pharmaceuticals, Wilmington MA, US).

Following the instructions of the SmPC, all lesions on the AMELUZ® side will be carefully wiped with an ethanol or isopropanol-soaked cotton pad to ensure degreasing of the skin. Scales and crusts will be removed accurately, and all lesion surfaces roughened gently. Care should be taken to avoid bleeding. AMELUZ® will be applied to the lesion area or the entire cancerized fields of about 20 cm2, using glove protected fingertips or a spatula. The gel should cover the lesions or entire fields and approximately 5 mm of the surrounding area with a film of about 1 mm thickness. The entire tube of AMELUZ® will be applied. The gel will be allowed to dry for approximately 10 minutes, before a light-tight dressing is placed over the treatment site. Following 3 hours of incubation, the dressing will be removed and the remnant gel wiped off .

Following the instructions of it's USPI, the LEVULAN® KERASTICK® topical solution is prepared by crushing the glass ampoules and mixing the contents together for at least 30 seconds. Following solution admixture, the cap from the LEVULAN® KERASTICK® applicator will be removed and the dry applicator tip should be dabbed on a gauze pad until uniformly wet with solution. Actinic keratoses targeted for treatment on the LEVULAN side should be clean and dry prior to applying the LEVULAN® KERASTICK® topical solution. The solution will be applied directly to the target lesions by dabbing gently with the wet applicator tip. Enough solution should be applied to uniformly wet the lesion surface, including the edges without excess running or dripping. The upper extremity shall be occluded with low density polyethylene plastic wrap and held in place with an elastic net dressing. The patient should wear a long-sleeved shirt and/or gloves or other protective apparel to shade the treated actinic keratoses from sunlight or other bright light sources until BLU-U® Blue Light Photodynamic Therapy Illuminator treatment. Photosensitization of the treated lesions will take place for 3 hours. The actinic keratoses should not be washed during this time. The occlusive dressing should be removed prior to light treatment and the treated area(s) gently rinsed with water and patted dry before light illumination.

Following the 3-hour incubation, the AMELUZ® treated side will be exposed to the BF-RhodoLED® lamp for 10 minutes to apply a light dose of 37 J/cm2 at 635 nm ± 9 nm. Simultaneously, the LEVULAN® KERASTICK® treated side will be exposed to the BLU-U® (Blue light photodynamic Therapy Illuminator Model 4170), for 16 minutes and 40 seconds to apply a light dose of approximately 10 J/cm2 at 417 nm ±5 nm.

Immediately following the illumination, subjects will grade the pain they experienced during treatment on a standard 11-point scale (none [0] to severe [10]; Appendix E). Subjects will be advised to avoid direct sunlight without application of sunscreen and exposure to intense lights such as tanning beds and sun lamps for 48 hours post-procedure.

Subjects will be visiting the office 60 days following PDT to assess the treatment areas. PDT will be repeated at this 60-day visit for any actinic keratosis lesions remaining in the treatment area. If a second PDT is performed, the subject will visit the office for the final assessment of the primary part of the study 60 days following the second treatment. Follow-up visits will occur at 6 months and 12 months following the last PDT treatment to determine recurrence rates.

Investigators will perform the following assessments:

1. Complete clearance of treated lesions.
2. Adverse Events (AEs): Post-procedure healing will be documented with investigator-rated standardized scales and assessment of adverse events post-treatment and at each follow-up visit post-treatment (Appendix A). Pain during illumination will be recorded comparing pain on both sides of the patient
3. Questionnaire

Subjects will perform the following self-assessments:

1. Subject Satisfaction: Subjects will assess satisfaction with treatment on a standardized 6-point scale (Appendix B) post-treatment and at each follow-up visit
2. Subject Pain Assessment: Pain during illumination will be assessed on both sides
3. Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Male or females ages 35-85
* Fitzpatrick skin type I through IV
* Participants with 4 to 17 clinically confirmed AK lesions of mild to moderate intensity according to Olsen grading in each of two comparable treatment fields on both hands or arms of the patients. The location and maximal size of the treatment fields should be such that PDT is possible with one illumination with BF-RhodoLED® and Blu-U® in parallel. The number of lesions on the two sides of a patient will not be allowed to differ by more than 50%
* Must be willing to give and sign a HIPPA form, photo consent and informed consent form °. Must be willing to comply with study dosing and complete the entire course of the study 6° Female patients will be either of non-childbearing potential defined as: A. Having no uterus B. No menses for at least 12 months with absence of other underlying cause C. (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as: Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device, Intrauterine coil, Bilateral tubal ligation, Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom), Abstinence (If practicing abstinence must agree to use barrier method described above (d) if becomes sexually active), Vasectomized partner D. Negative urine pregnancy test results Baseline prior to study entry, Day 30, and Day 60

Exclusion Criteria:

* Hypersensitivity to porphyrins.
* Known hypersensitivity to study medication, which includes soybean phosphatidylcholine.
* Diagnosis of porphyria or photodermatoses.
* Use of photosensitizing medications such as St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones, and tetracyclines within 1 month of study initiation.
* Presence of wound, suspected BCC or SCC, scar or tattoo, or co-existing potentially confounding skin condition within treatment area.
* Previous PDT in the treatment area within the past 6 months.
* Use of oral/topical retinoids within the treatment area within 1 month of baseline.
* Subjects with recently excessive exposure of the treatment area to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study.
* Female subjects who are pregnant, nursing an infant or planning a pregnancy during the study throughout the course of the study.
* Presence or evidence of any conditions that in the opinion of the investigator might impede the subject's ability to give consent or comply with protocol requirements.
* Ablative laser resurfacing to on their upper extremities within 12 months.
* Non-ablative laser or light procedures to their upper extremities within the past 3 months.
* Microdermabrasion (light or medium skin peel) treatment on their upper extremities within the past 30 days.
* Subjects who have participated in another clinical trial within the past 30 days.
* Presence of any physical conditions which, in the opinion of the investigator, may create an additional risk to subject safety or compromise their ability to comply with the study protocol.
* Presence of any psychological conditions or use of medications which may compromise a subject's ability to comply with the study protocol or provide informed consent
* History of non-compliance with previous clinical trial protocols.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Total Lesion Clearance Rate | Baseline to Month12 Post Final PDT
  Percent change in number of lesions on each treatment side

SECONDARY OUTCOMES:
Cosmetic Outcome | Baseline to Month12 Post Final PDT
  Cosmetic changes as assessed by Investigator
Subject Satisfaction | Baseline to Month12 Post Final PDT
  Subject Self Assessment of Satisfaction where 1 = Extremely Satisfied, 2 = Satisfied, 3 = Slightly Satisfied, 4 = Slightly Dissatisfied, 5 = Dissatisfied, 6 = Extremely Dissatisfied
Clinical Recurrence | Month12 Post Final PDT
  Investigator Assessed Recurrence of Treated AKs

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmetic Laser Dermatology/West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No